CLINICAL TRIAL: NCT03378830
Title: Pain at Home After Tonsillectomy With or Without Adenoidectomy
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Karen Brown, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2017-3127
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Sleep Apnea; Adenotonsillectomy; Pediatric ALL
Keywords: Pain; Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study type is a prospective observational cohort study of children undergoing adenotonsillectomy (T&A). The study will recruit the annual caseload of children undergoing T&A at the Montreal Children's Hospital, QC, Canada; aiming for 200 children. There are no interventions.

The purpose of this study is to determine the severity and duration of postoperative pain after T&A and to link the severity of this pain with the severity of sleep disordered breathing.

DETAILED DESCRIPTION:
Adenotonsillectomy (T&A) is one or the most common surgeries performed in children. Even though T&A is considered a painful surgery, it is often scheduled as a day surgery and parents manage the postoperative pain at home. Historically, the home analgesic following adenotonsillectomy consisted of a combination of acetaminophen and codeine. In June 2013, Health Canada no longer recommended the use of codeine in children less than 12 years of age. Thus in current practice the discharge analgesic is a combination of ibuprofen, acetaminophen and oral rescue morphine. This shift in practice has occurred globally as well as in our institution without evaluating the impact on analgesia at home following T&A.

The published literature reports that as many as 50% of children managed with the acetaminophen/codeine regimen visit a primary care physician for the management of pain/infection following T&A and a high proportion of these children are prescribed an opioid. This practice is of concern for the following reasons. Sleep disordered breathing (SDB) is the most common indication for T&A in children. In some children the sleep disturbance meets the diagnostic criteria for obstructive sleep apnea (OSA). A subset of children, with severe OSA are more sensitive to both the analgesic and respiratory effects of opioids. In these children, an age-appropriate dose of opioids may result in an overdose.

Study Design:

Pain will be measured in hospital and at home with validated pain scores. The primary outcome measure is the Parents' Postoperative Pain Measure (PPPM), a valildated, established metric, with good construct and content validity, for the repeated evaluation of pain following surgery in the home environment. Parents will be asked to record the both the pain scores, twice daily for 14 days.

A secondary outcome measure will be the self report of pain from the children. Two validated pain scales will be used. For pre-verbal children, the Face, Legs, Activity, Cry and Consolability (FLACC) pain scale will be used. This 0-10 scale has shown good reliability, validity and relevance in clinical practice for children's less than 4 years of age for post-operative pain. For older children the modified modified Faces Pain Scale (FPS-R) will be used. The 0-10 metric score is validated and reliable for children aged 4 - 16 years.

Outcome measure Time Frame Parents will be asked to record the PPPM and either the FLACC or the FPS-R, twice daily for 14 days in a pain diary. The change in pain scores over 14 days will be evaluated.

Preoperatively the severity of the SDB will be assessed, with the Snoring, Trouble Breathing, UnRefreshed (STBUR) questionnaire; a 5-item questionnaire.

Primary Aim:

1) To determine the severity and duration of postoperative pain after adenotonsillectomy (T&A) and to correlate the pain scores with the STBUR.

ELIGIBILITY:
Inclusion Criteria:

* Elective scheduled surgery for adenotonsillectomy
* Fluency in French
* Fluency in English

Exclusion Criteria:

* Neuromuscular disease
* Seizure disorders,
* Cyanotic heart disease,
* Trisomy 21,
* Craniofacial syndromes such as Crouzons syndrome,
* Steroid dependant asthma,
* Cystic fibrosis,
* Bronchopulmonary dysplasia
* Severe autism .
* Developmental delay which impair the assessment of pain.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Otherwise healthy children aged 2 to 12 years I am not sure what the required sampling method means so I put non-probability sample.-
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Parent Pain Measure (PPPM) | We are asking the parents to record the PPPM twice daily for 14 days.
  The PPPM is a validated 15 item questionnaire that requires a Yes or No response. The maximum total score is 15. A total score above 6 indicates clinically relevant pain.

OTHER OUTCOMES:
The STBUR (Snoring, Trouble Breathing, UnRefreshed) questionnaire. | The STBUR will be administered once during the preoperative evaluation of the child.
  The STBUR is a 5 item questionnaire that requires a yes or no response. The STBUR has been validated to predict 1) perioperative respiratory adverse events and 2) opioid related respiratory adverse event. The maximum score is 5. A total score of 3 or more is associated with in increased risk of respiratory adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Brown, MD, Principal Investigator — Pediatric Anesthesiologist
Locations (1):
- The Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frigon C, Agnihotram RV, Berard-Giasson A, Lamonde F, Pang M, Daniel SJ, Brown KA. Association between obstructive sleep-disordered breathing severity and pain trajectories after adenotonsillectomy in children: a prospective cohort study. Br J Anaesth. 2026 Jan;136(1):167-178. doi: 10.1016/j.bja.2025.09.015. Epub 2025 Nov 28. PMID 41314942
- [Derived] Lima LACN, Otis A, Balram S, Giasson AB, Carnevale FA, Frigon C, Brown KA. Parents' perspective on recovery at home following adenotonsillectomy: a prospective single-centre qualitative analysis. Can J Anaesth. 2023 Jul;70(7):1202-1215. doi: 10.1007/s12630-023-02479-2. Epub 2023 May 9. PMID 37160822